CLINICAL TRIAL: NCT04883970
Title: CLDN18.2 Targeting 124I-18B10(10L) PET Imaging in Patients With Gastrointestinal Tumors
Brief Title: CLDN18.2 Targeting PET Imaging in Patients With Gastrointestinal Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021KT57
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Experimental): All study participants will be allocated to this arm (single-arm study). Study participants will undergo 124I-18B10(10L) PET/CT scans
  Interventions: Other: 124I-18B10(10L) PET/CT

INTERVENTIONS:
Other: 124I-18B10(10L) PET/CT — Study participants will undergo 124I-18B10(10L) PET/CT scans

SUMMARY:
The objective of the study is to constrcut a noninvasive approach 124I-18B10(10L) PET/CT to detect the CLDN18.2 expression of tumor lesions in patients with gastrointestinal tumors and to identify patients benefiting from CLDN18.2 targeting treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged >18 years old; ECOG 0 or 1;
* 2. Patients with Gastrointestinal tumors;
* 3. Has at least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST V1.1);
* 4. life expectancy >=12 weeks.

Exclusion Criteria:

* 1. Significant hepatic or renal dysfunction;
* 2. Is pregnant or ready to pregnant;
* 3. Cannot keep their states for half an hour;
* 4. Refusal to join the clinical study;
* 5. Suffering from claustrophobia or other mental diseases;
* 6. Any other situation that researchers think it is not suitable to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- HUA ZHU, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang S, Qi C, Ding J, Li D, Zhang M, Ji C, Jiang F, Teng F, Yu J, Qian X, Wang F, Shen L, Gao J, Yang Z, Zhang C, Zhu H. First-in-human CLDN18.2 functional diagnostic pet imaging of digestive system neoplasms enables whole-body target mapping and lesion detection. Eur J Nucl Med Mol Imaging. 2023 Jul;50(9):2802-2817. doi: 10.1007/s00259-023-06234-z. Epub 2023 Apr 26. PMID 37099132